CLINICAL TRIAL: NCT00195091
Title: A Phase II Study of Tetrathiomolybdate (TM) in Patients With Breast Cancer at Moderate to High Risk of Recurrence
Brief Title: Phase II Study of Tetrathiomolybdate (TM) in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left MSKCC
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-023; 0309006307 (Other: Weill Cornell Medical College)
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2024-04-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tetrathiomolybdate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tetrathiomolybdate (TM) (Experimental): Induction period - TM 40 mg is administered three x per day with meals and TM 60 mg at bedtime for a total of 4 doses (180 mg) per day.
  Maintenance Period - Total TM dose per day will be in 20 mg increments to tailor the therapy to individualized patient needs to maintain the Cp level at 5-17mg/dL. Thus all dose modifications will be dependent on individual patient Cp levels. TM 40 mg p.o. BID with meals and TM 20 mg at bedtime. Subjects who have no evidence of disease (NED) and are receiving a benefit of TM can continue taking the drug for up to 120 months.
  Interventions: Drug: Tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate — Induction with Tetrathiomolybdate (TM) Tetrathiomolybdate 40 mg. p.o. TID with meals and tetrathiomolybdate 60 mg at bedtime for a total of 4 doses (180 mg) per day.
  Induction goal Total tetrathiomolybdate dose per day = 180 mg until serum ceruloplasmin (Cp) level decreases to 5-15mg/dL.
  When target Cp window is reached, then the maintenance phase begins.
  Maintenance with Tetrathiomolybdate Total tetrathiomolybdate dose per day = 100 mg
  Tetrathiomolybdate 40 mg p.o. BID with meals and tetrathiomolybdate 20 mg at bedtime.
  Other Names: TM

SUMMARY:
Patients with moderate to high risk primary breast cancer (Stage II with more than 4 lymph nodes involved with cancer) III or Stage IV (without evidence of disease) will take tetrathiomolybdate (TM) pills for two years.

The objectives of the study are to:

* Assess the safety and tolerability of tetrathiomolybdate in patients with breast cancer at high risk of tumor recurrence.
* Observe the disease-free survival of patients in this trial.
* Conduct background scientific experiments on tumor tissue and blood of patients in this study

DETAILED DESCRIPTION:
Patients with moderate to high risk primary breast cancer -Stage III, Triple negative (T= 4 cm N0, any N+), Stage IV (without evidence of disease) will take tetrathiomolydbate (TM) pills for two years.

Extension study 1 - If patients are shown to be copper depleted, they are given the option to continue to receive TM for an additional 2 years.

Extension study 2 - Open to patients who are stage 4 NED, 10 involved lymph nodes or triple negative molecular subtype and candidates will continue for months 49-72.

Extension study 3 - Open to patients who are stage 4 NED receiving a benefit from TM. These subjects can continue receiving TM for 73-96 months.

Extension study 4 - Open to patients who are stage 4 NED receiving a benefit from TM. These subject can continue receiving TM for 97-120 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed breast malignancy that is:

   * High risk stage II breast cancer (≥4 positive lymph nodes),
   * Stage III breast cancer, including inflammatory breast cancer
   * Stage IV breast cancer in a complete remission (bone only not allowed unless the bone scan is normal).
2. The patient must have had what is considered standard adjuvant systemic therapy that may include chemotherapy, hormonal therapy and radiation therapy. They may have undergone high dose chemotherapy with stem cell support as part of their therapy in the adjuvant or metastatic setting. The patient is allowed to continue to take adjuvant hormonal therapy (for high risk adjuvant patients) and may be allowed to be on hormonal consolidation post transplant if they are without evidence of disease after a transplant for metastatic breast cancer. The patient cannot be actively receiving chemotherapy or any biologic agent to treat their breast cancer.
3. Six weeks must elapse from last chemotherapy or radiation therapy.
4. The patient must have had definitive surgical therapy for their breast cancer. This includes lumpectomy and axillary dissection or mastectomy.
5. No clinical or radiologic evidence of disease after surgery and/or systemic treatment (by CT scan of chest, abdomen and pelvis and bone scan or PET scan prior to enrollment)
6. Because no dosing or adverse event data are currently available on the use of TM in patients < 18 years of age, children are excluded from this study.
7. ECOG performance status < 1
8. Life expectancy of greater than 3 months.
9. Patients must have normal organ and marrow function as defined below:

   * hemoglobin >10mg/dL
   * absolute neutrophil count >1,500/mL
   * platelets >100,000/mL
   * total bilirubin < 1.5 x normal institutional limits
   * AST(SGOT)/ALT(SGPT) <1.5 X institutional upper limit of normal
10. Erythropoietin alpha is allowed, as indicated.
11. Bisphosphonates may be administered if they were started prior to starting this therapy.
12. Patients must be on stable medical therapy for at least 2 weeks if they are being treated medically for their peripheral neuropathy.
13. Concurrent herceptin is not allowed.
14. The effects of TM on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
15. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 6 weeks prior to entering the study.
2. Objective evidence of breast cancer.
3. Carcinomatous meningitis or history of neoplastic parenchymal brain disease.
4. Serum creatinine >1.5 x normal.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TM.
6. Pregnant women are excluded from this study because TM has the potential to have teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TM, breastfeeding should be discontinued if the mother is treated with TM.
7. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with TM.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-12; Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vahdat, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Ramchandani D, Berisa M, Tavarez DA, Li Z, Miele M, Bai Y, Lee SB, Ban Y, Dephoure N, Hendrickson RC, Cloonan SM, Gao D, Cross JR, Vahdat LT, Mittal V. Copper depletion modulates mitochondrial oxidative phosphorylation to impair triple negative breast cancer metastasis. Nat Commun. 2021 Dec 15;12(1):7311. doi: 10.1038/s41467-021-27559-z. PMID 34911956
- See also: Related Info — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a transfer study from Weill Cornell to MSKCC. Participants were consented at Weill Cornell and transferred to MSKCC.
Groups:
- Tetrathiomolybdate (TM): Tetrathiomolybdate: Induction with Tetrathiomolybdate (TM)
  When target Cp window is reached, then the maintenance phase begins.
Period: Overall Study
Arm/Group | Tetrathiomolybdate (TM)
Started | 16
Completed | 0
Not Completed | 16
Not completed — Study terminated and PI has left MSKCC | 16

BASELINE CHARACTERISTICS:
Arm/Group | Tetrathiomolybdate (TM)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 64 [51 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression for Patients With Breast Cancer Treated With Study Drug
Time Frame: duration of study
Population: N/A - data were not collected
Arm/Group | Tetrathiomolybdate (TM)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tetrathiomolybdate (TM)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT00195091/Prot_SAP_000.pdf